CLINICAL TRIAL: NCT05496335
Title: A Phase 1 Study to Evaluate Sequential Administration of AGN-151586 and OnabotulinumtoxinA (BOTOX) in Subjects for Treatment of Glabellar Lines
Brief Title: A Study to Evaluate Sequential Administration of AGN-151586 and OnabotulinumtoxinA (BOTOX) Injections in Adult Participants for Treatment of Glabellar Lines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M23-365
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Glabellar Lines
Keywords: AGN-151586; OnabotulinumtoxinA; BOTOX
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- AGN-151586, BOTOX (Experimental): Participants will receive 5 intramuscular injections of AGN-151586 in the glabellar complex on Day 1. Eligible participants will receive BOTOX injections and will be followed for up to 4 months.
  Interventions: Drug: AGN-151586; Drug: BOTOX
- Placebo, BOTOX (Experimental): Participants will receive 5 intramuscular injections of placebo in the glabellar complex on Day 1. Eligible participants will receive BOTOX injections and will be followed for up to 4 months.
  Interventions: Drug: BOTOX; Drug: Placebo

INTERVENTIONS:
Drug: AGN-151586 — Intramuscular Injection
  Arms: AGN-151586, BOTOX
Drug: BOTOX — Intramuscular Injection
  Other Names: OnabotulinumtoxinA
Drug: Placebo — Intramuscular Injection
  Arms: Placebo, BOTOX

SUMMARY:
Facial lines that develop from repeated facial expression, such as glabellar lines (GL), are typically treated by selectively weakening specific muscles with small quantities of botulinum toxin. The purpose of this study is to assess how safe and effective sequential administration of AGN-151586 and OnabotulinumtoxinA (BOTOX) is in adult participants with moderate to severe GL.

AGN-151586 is an investigational product being developed for the treatment of GL. Participants are placed in 1 of 2 groups, called treatment arms. Each group receives a different treatment. One group will receive AGN-151586 followed by BOTOX and the other group will receive placebo followed by BOTOX. There is a 1 in 2 chance that participants will be assigned to placebo. Around 80 adult participants with moderate to severe GL will be enrolled in the study in approximately 10 sites around the United States.

Participants will receive either AGN-151586 or Placebo administered as 5 intramuscular injections to the glabellar complex on Day 1. Eligible participants may then receive BOTOX injections on Day 30 and will be followed for up to 4 months.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to accurately assess their facial lines without the use of eyeglasses (contact lens use is acceptable).
* Participants with moderate or severe Glabellar Lines at maximum frown as assessed by both the investigator and participant using the Facial Wrinkle Scale (FWS) at screening and baseline (Day 1) visit.

Exclusion Criteria:

* Uncontrolled systemic disease.
* Presence or history of any medical condition that may place the participant at increased risk following exposure to AGN-151586 or BOTOX interfere with the study evaluation, including:

  * Diagnosed myasthenia gravis, Lambert-Eaton syndrome, amyotrophic lateral sclerosis, or any other significant disease that might interfere with neuromuscular function
  * History of facial nerve palsy
  * Infection or dermatological condition at the treatment injection sites
  * Marked facial asymmetry, dermatochalasis, deep dermal scarring, excessively thick sebaceous skin, excessively photodamaged skin, or the inability to substantially lessen facial lines even by physically spreading them apart
  * Any eyebrow or eyelid ptosis at screening or Baseline Day 1 visit as determined by the investigator
* History of clinically significant drug, nicotine, or alcohol abuse within the last 6 months.
* Tattoos, jewelry, or clothing which obscure the glabellar area and cannot be removed.
* History of known immunization to any botulinum neurotoxin serotype.
* Anticipated need for surgery or overnight hospitalization during the study.
* History of surgical procedures on forehead and/or periorbital areas or affecting these areas including any lifting procedure (e.g., rhinoplasty, facial lift, suture lift, thread lift, brow lift, eyelid and/or eyebrow surgery).
* History of periorbital, mid-facial, or upper-facial treatment with semi permanent or permanent soft tissue fillers (e.g., poly-L-lactic acid, polyalkylimide, polymethylmethacrylate, polytetrafluoroethylene, and silicone), synthetic implantation and/or autologous fat transplantation.
* Known active severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection or participants with a positive polymerase chain reaction (PCR) test in the past 14 days prior to Baseline Day 1 who are asymptomatic.
* Participant who has been treated with any investigational drug within 30 days or 5 half-lives of the drug (whichever is longer) prior to the first dose of study drug or is currently enrolled in another clinical study or was previously enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants achieving "none" or "mild" on the Facial Wrinkle Scale (FWS) according to the investigator assessment of Glabellar Lines (GL) severity at maximum frown | At Day 60
  The investigator assessment of GL severity at maximum frown using a 4-grade scale (0 to 3) where 0=none and 3=severe.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (10):
- United States (10):
  - The Eye Research Foundation /ID# 244430, Newport Beach, California
  - Cosmetic Laser Dermatology /ID# 244425, San Diego, California
  - AboutSkin Research, LLC /ID# 244416, Greenwood Village, Colorado
  - Skin Research Institute LLC /ID# 244424, Coral Gables, Florida
  - Skin and Cancer Associates, LLP /ID# 244415, Miami, Florida
  - DeNova Research /ID# 244421, Chicago, Illinois
  - Advanced Dermatology /ID# 244427, Lincolnshire, Illinois
  - Laser and Skin Surgery Center of Indiana /ID# 244423, Indianapolis, Indiana
  - Bellaire Dermatology Associates /ID# 244428, Bellaire, Texas
  - Premier Clinical Research /ID# 244429, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No